CLINICAL TRIAL: NCT05206474
Title: Open, Non-comparative, Multicentre Clinical Investigation to Evaluate the Performance and Safety of the Medical Device IRADYN® (Polymerized Polynucleotides) Intra-articularly Administered in Subjects With Osteoarthritis of the Knee
Brief Title: To Evaluate the Performance and Safety of the Medical Device IRADYN in Subjects With Osteoarthritis of the Knee
Acronym: IRADYN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: I.R.A. Istituto Ricerche Applicate S.p.A. (Network)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPIRA/0121/MD
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Joint Inflammation; Iradyn; Polynucleotides; Filler
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis

STUDY DESIGN:
Intervention Model Description: Open-Label, non-comparative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IRADYN (Experimental): One group, all patients will receive IRADYN® (intra-articular administration).
  One course of IRADYN® at baseline, consisting of a mono-dose intra-articular administration (2ml).
  From week 1 to week 6, injection will be performed, if necessary, during the visit, following the dosage reported in the instruction for use / summary of product characteristic.
  Interventions: Device: IRADYN

INTERVENTIONS:
Device: IRADYN — One course of IRADYN® at baseline, consisting of a mono-dose intra-articular administration (2 ml).
  From week 1 to week 6, injection will be performed, if necessary, during the visit, following the dosage reported in the instruction for use / summary of product characteristic.

SUMMARY:
The benefits of single or repetitive administration (1 to 6) can have similar result in terms of muscular strength and patients' quality of life improvement, benefiting of the advantages of polymerized polynucleotides (IRADYN) formulation.

DETAILED DESCRIPTION:
Of all osteoarthritis' localization into human body, knee OA represents the most common OA localization.

On 2014 the European Society for Clinical and Economic Aspects of Osteoporosis and Osteoarthritis (ESCEO) has suggested as first step of pharmacological treatment for knee osteoarthritis (OA) a background therapy with chronic symptomatic slow-acting drugs for osteoarthritis (SYSADOAs). In this class of natural compounds, hyaluronic acid (HA) has evidenced its efficacy after intra-articular (IA) administration in patient with mild to moderate knee OA .

The filler used in this clinical investigation is using polymerised polynucleotides (PDRN) that has hydrophilic properties of polyanions; therefore, it can bind water molecules and provide a moisturising and lubricant effect. Its viscoelastic properties allow it to compensate for the loss of synovial fluid viscosity in the event of degenerative or trauma joint alterations. These actions reduce the mechanical stress on joints, thereby decreasing friction. This improves joint function and movement with significant relief of pain commonly associated with this problem. Moreover, the enzymatic degradation of the polynucleotide chain releases nucleotides into the synovial cavity. These nucleotides can bind water molecules and share the same viscoelastic properties as the entire chain, helping extend the duration of the effect.

The benefits of single or repetitive administration (1 to 6) can have similar result in terms of muscular strength and patients' quality of life improvement, benefiting of the advantages of polymerized polynucleotides (IRADYN) formulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 80 years (inclusive, ≥ 40 and ≤ 80 years);
* Symptomatic knee osteoarthritis as defined by the American College of Rheumatology (ACR) criteria (for subjects with OA at both knees, the most painful one will be included in the study only, respecting Kellgren-Lowrance grade II or III);
* Ambulant without assistance;
* Kellgren-Lawrence grade II or III on X-ray performed at maximum 6 months before screening;
* Visual Analogue Scale (VAS) score knee pain ≥40 at screening and 30 days before;
* Oral/parenteral corticosteroid or NSAIDs (≤10 mg prednisone) administration at least 30 days before screening.
* Signed Informed consent

Exclusion Criteria:

* Unstable knee;
* Varus or valgus ≥ 15 degrees;
* Active malignancy;
* Knee trauma or lose body parts 1 year before screening;
* Rheumatoid Arthritis, avascular necrosis, fibromyalgia;
* Use of potent analgesics 15 days (different from ≤ 10 mg prednisone) before screening;
* Intra-articular HA, polymerized polynucleotides or corticosteroid injection within 6 months before screening;
* Arthroscopic or knee open surgery within 12 months before screening;
* Body Mass Index (BMI) ≥ 40 kg/m2;
* Active infection around the injection site;
* Use of anticoagulants or history of thrombocytopenia;
* Concomitant use of disease-modifying antirheumatic drugs (DMARDs), anaesthetics;
* Known sensitivity to polymerized polynucleotides;
* Pregnancy, breast feeding.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-07 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Range of Motion (ROM) | 14 weeks compared with baseline
  Change in Range of Motion (ROM) parameters, measured in degrees, using a goniometer (Active Knee Flexion - AKF, Passive Knee Flexion - PKF, Active Knee Extension - AKE, Passive Knee Extension - PKE)
Change in Visual Analogue Scale (VAS) for pain (at rest) | 14 weeks compared to baseline
  Visual Analogue Scale (VAS) for pain at rest is a 100 mm chart-line scale for the mentioned situation on which the subject must draw a mark on the scale to emphasize the intensity of the pain.
  Minimum score is 0 and it means no pain. Maximum score is 100 and represents the maximum pain that patient can suffer.

SECONDARY OUTCOMES:
Absolute change in Visual Analogue Scale (VAS) for pain (on moving and on pressing) | Up to 14 weeks
  Absolute change in VAS for pain (on moving and on pressing) at all visits compared to Baseline Visit. Visual Analogue Scale (VAS) for pain under pressure and at movement is a 100 mm chart-line scale for each of the mentioned situations on which the subject must draw a mark on the scale to emphasize the intensity of the pain.
  Minimum score is 0 and it means no pain. Maximum score is 100 and represents the maximum pain that patient can suffer.
Absolute change in Knee injury and Osteoarthritis Outcome Score (KOOS) | 6 weeks and 14 weeks compared to baseline
  KOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Physician Efficacy Global Evaluation | 14 weeks
  Percentage of patients with "very good efficacy" evaluations in the Physician Efficacy Global Evaluation assessed at week 14.
Evaluation of NSAIDs consumption at all visits | up to 14 weeks
  Incidence of Non-steroidal anti-inflammatory drugs (NSAIDs) consumption from first visit to final visit.

OTHER OUTCOMES:
AE, SAE, ADE, SADE, DD incidence | 14 weeks
  Adverse Event, Serious Adverse events, Adverse Device Event, Serious Adverse Device Event, Device Deficiency incidence
Patient Global Tolerability | 14 weeks
  Percentage of patients with "very good" evaluations in the Patient Global Tolerability assessed at all visits.

CONTACTS AND LOCATIONS:
Overall Officials: George Puenea, MD, Principal Investigator — Fizio Center
Locations (2):
- Romania (2):
  - Centrul de kinetoterapie si Masaj Banat, Timișoara, Timiș County
  - Fizio Center, Timișoara, Timiș County